CLINICAL TRIAL: NCT04506307
Title: Noninvasive Fat Reduction With the CoolSculpting System
Brief Title: CoolSculpting System
Acronym: ELI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeltiq Aesthetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ZA20-001
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Body Fat Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fat Reduction (Experimental): The treatments are designed to see if the fat can be reduced in the torso area with a new applicator design.
  Interventions: Device: The ZELTIQ System

INTERVENTIONS:
Device: The ZELTIQ System — The CoolSculpting machine will be used to perform the treatments.

SUMMARY:
Evaluate the safety and efficacy of multiple, simultaneous CoolSculpting cycles for the purpose of non-invasive fat reduction.

ELIGIBILITY:
Inclusion Criteria

* Subject (healthy volunteer) has read and signed the study written informed consent form.
* Male or female ≥ 22 years and ≤65 years of age.
* Subject has clearly visible fat in one or more areas on the torso (abdomen, flank, back fat, bra fat), which in the investigator's opinion, may benefit from the treatment.
* Subject has not had weight change exceeding 5% of body weight in the preceding month.
* Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the study.
* Subject has a BMI ≤ 30 as determined at screening.
* Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

Exclusion Criteria

* Subject has had a recent surgical procedure in the area of intended treatment.
* Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
* Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
* Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
* Subject has a known history of cryoglobulinemia, paroxysmal cold hemoglobinuria, or cold agglutinin disease.
* Subject has a known sensitivity to cold, such as cold urticaria, Raynaud's disease, chilblains (pernio), or any known condition with a response to cold exposure that limits blood flow to the skin.
* Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
* Subject is taking or has taken diet pills or supplements within the past month.
* Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
* Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
* Subject has a history of hernia in the area(s) to be treated.
* Subject is pregnant or intending to become pregnant during the study period (in the next 8 months).
* Subject is lactating or has been lactating in the past 6 months.
* Subject is unable or unwilling to comply with the study requirements.
* Subject is currently enrolled in a clinical study of any unapproved investigational drug or device.
* Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-03-13 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-10-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Zeltiq Aesthetics
Locations (4):
- United States (4):
  - Marina Plastic Surgery, Marina del Rey, California
  - Leyda E Bowes MD, Pleasanton, California
  - Moradi MD Cosmetic Surgery, Vista, California
  - Riverchase Dermatology, Miami, Florida

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CoolSculpting of the Torso: Participants were to receive 2 CoolSculpting treatments of the torso (abdomen, flanks, bra fat, and/or back fat) performed at 6 weeks apart.
Period: Overall Study
Arm/Group | CoolSculpting of the Torso
Started | 35
Received 1 Treatment | 35
Received 2 Treatments | 30
Completed | 33
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least 1 treatment.
Arm/Group | CoolSculpting of the Torso
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 1
  Race: Asian | 4
  Race: Black or African American | 2
  Race: White | 24
  Race: Other | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Photographs Correctly Identified by At Least 2 of 3 Blinded Reviewers From the Independent Physician Reviewer Panel
Description: Photographs of the treatment areas (torso) taken at baseline and 12-weeks after final treatment were assessed by blinded independent reviewers to determine if the CoolSculpting treatment had the effect of improvement in the reduction of fat. The reviewers were presented with 2 series of photographs the baseline and the post final treatment series, and asked to select the series representing the baseline photographs. The order in which the photographs were presented was randomized by participant. Reported here is the percentage (%) of images that were correctly identified by at least 2 out of 3 blinded independent reviewers. Success was defined as at least 70% correct identification of the baseline images.
Time Frame: Week 12 post final treatment (18 weeks after first treatment)
Population: Per Protocol population consisted of participants who received 2 treatments and had a weight change of no more than 5% of total body weight at the time the 12-week assessments were performed compared to the weight obtained at the first treatment visit. In addition, participants with extensive tattoos in the treated area that could hinder the evaluation were excluded.
Measure: Number (95% Confidence Interval); unit: % of images identified correctly
Arm/Group | CoolSculpting of the Torso
Number analyzed (Participants) | 28
% of images identified correctly | 75.0 [55.1 to 89.3]

2. Secondary Outcome: Number of Participants With Device and/or Procedure Related Adverse Events (AEs) and Device-related Serious Adverse Events (SADEs)
Description: An AE was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in participants, whether or not considered related to treatment. A serious adverse event (SAE) was an AE that resulted in death, serious deterioration in health, permanent impairment of a body structure/function, was life-threatening, required hospitalization or medical/surgical intervention, led to fetal distress or death, congenital abnormality, or birth defect. An ADE was any sign, symptom, or disease that was determined by the Investigator to have a causal relationship or possible causal relationship with the investigational device, including any AE resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the device or from use error or intentional misuse of the device. A SADE was an ADE that resulted in any of the consequences characteristic of an SAE.
Time Frame: From first treatment up to Week 12 post final treatment (18 weeks after first treatment)
Population: The Safety Population consisted of all enrolled participants who received at least 1 treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | CoolSculpting of the Torso
Number analyzed (Participants) | 35
Participants
  Device and/or Procedure Related AEs | 11
  SADEs | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 12 weeks post final treatment (up to 18 weeks)
Description: The Safety Population consisted of all enrolled participants who received at least 1 treatment.
Arm/Group | CoolSculpting of the Torso
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 11/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CoolSculpting of the Torso (N=35)
Urinary tract infection (Infections and infestations) | 1
Back injury (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CoolSculpting of the Torso (N=35)
COVID-19 (Infections and infestations) | 2
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2
Vasovagal event (General disorders) | 4
Subcutaneous induration (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-19): https://cdn.clinicaltrials.gov/large-docs/07/NCT04506307/Prot_SAP_000.pdf